CLINICAL TRIAL: NCT01189240
Title: Phase I/II Study of R04929097 With Bevacizumab in Patients With Recurrent Malignant Glioma
Brief Title: RO4929097and Bevacizumab in Treating Patients With Progressive or Recurrent Malignant Glioma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Company decided to stop development of drug - 7/31/12
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2011-02509; NCI-2011-02509 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000683099; ABTC-1002 (Other: Adult Brain Tumor Consortium); ABTC-1002 (Other: CTEP); U01CA137443 (NIH)
Record Dates: First submitted 2010-08-25; First posted 2010-08-26 (Estimated); Results first posted 2015-07-14 (Estimated); Last update posted 2015-12-14 (Estimated); Status verified 2015-10

CONDITIONS: Adult Anaplastic Astrocytoma; Adult Anaplastic Oligodendroglioma; Adult Giant Cell Glioblastoma; Adult Glioblastoma; Adult Gliosarcoma; Recurrent Adult Brain Tumor
MeSH Terms: conditions — Astrocytoma; Oligodendroglioma; Glioblastoma; Gliosarcoma; Brain Neoplasms | interventions — 2,2-dimethyl-N-(6-oxo-6,7-dihydro-5H-dibenzo(b,d)azepin-7-yl)-N'-(2,2,3,3,3-pentafluoropropyl)malonamide; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (7):
- Phase I Dose Finding (Experimental): Patients receive oral gamma-secretase/Notch signalling pathway inhibitor RO49290977 on days 1-3, 8-10, 15-17, and 22-24, and bevacizumab IV over 30-90 minutes on days 1 and 15. Other: pharmacological study: correlative studies; laboratory biomarker analysis: correlative studies.
  Interventions: Drug: gamma-secretase/Notch signalling pathway inhibitor RO4929097; Biological: bevacizumab; Other: laboratory biomarker analysis; Other: pharmacological study
- Phase II Stage I (Experimental): Patients receive oral gamma-secretase/Notch signalling pathway inhibitor RO49290977 on days 1-3, 8-10, 15-17, and 22-24, and bevacizumab IV over 30-90 minutes on days 1 and 15.Other: laboratory biomarker analysis: correlative studies.
  Phase 2 - not implemented due to drug supply from company
  Interventions: Drug: gamma-secretase/Notch signalling pathway inhibitor RO4929097; Biological: bevacizumab; Other: laboratory biomarker analysis
- Phase II Stage II Arm 1 (Experimental): Patients receive oral gamma-secretase/Notch signalling pathway inhibitor RO49290977 on days 1-3, 8-10, 15-17, and 22-24, and bevacizumab IV over 30-90 minutes on days 1 and 15. Other: laboratory biomarker analysis: correlative studies.
  Phase 2 - not implemented due to drug supply from company
  Interventions: Drug: gamma-secretase/Notch signalling pathway inhibitor RO4929097; Biological: bevacizumab; Other: laboratory biomarker analysis
- Phase II Stage II Arm 2 (Active Comparator): Patients receive bevacizumab IV over 30-90 minutes on days 1 and 15. Other: laboratory biomarker analysis: correlative studies.
  Phase 2 - not implemented due to drug supply from company
  Interventions: Biological: bevacizumab; Other: laboratory biomarker analysis
- Phase I Dose Finding - Level 1 5mg (Experimental): Patients receive oral gamma-secretase/Notch signalling pathway inhibitor RO49290977 5mg on days 1-3, 8-10, 15-17, and 22-24, and bevacizumab IV over 30-90 minutes on days 1 and 15. Other: pharmacological study: correlative studies; laboratory biomarker analysis: correlative studies.
  Interventions: Drug: gamma-secretase/Notch signalling pathway inhibitor RO4929097; Biological: bevacizumab; Other: laboratory biomarker analysis; Other: pharmacological study
- Phase I Dose Finding - Level 2 10mg (Experimental): Patients receive oral gamma-secretase/Notch signalling pathway inhibitor RO49290977 10mg on days 1-3, 8-10, 15-17, and 22-24, and bevacizumab IV over 30-90 minutes on days 1 and 15. Other: pharmacological study: correlative studies; laboratory biomarker analysis: correlative studies.
  Interventions: Drug: gamma-secretase/Notch signalling pathway inhibitor RO4929097; Biological: bevacizumab; Other: laboratory biomarker analysis; Other: pharmacological study
- Phase I Dose Finding - Level 3 20mg (Experimental): Patients receive oral gamma-secretase/Notch signalling pathway inhibitor RO49290977 20mg on days 1-3, 8-10, 15-17, and 22-24, and bevacizumab IV over 30-90 minutes on days 1 and 15. Other: pharmacological study: correlative studies; laboratory biomarker analysis: correlative studies.
  Interventions: Drug: gamma-secretase/Notch signalling pathway inhibitor RO4929097; Biological: bevacizumab; Other: laboratory biomarker analysis; Other: pharmacological study

INTERVENTIONS:
Drug: gamma-secretase/Notch signalling pathway inhibitor RO4929097 — Given orally
  Other Names: R4733; RO4929097
  Arms: Phase I Dose Finding; Phase I Dose Finding - Level 1 5mg; Phase I Dose Finding - Level 2 10mg; Phase I Dose Finding - Level 3 20mg; Phase II Stage I; Phase II Stage II Arm 1
Biological: bevacizumab — Given IV
  Other Names: anti-VEGF humanized monoclonal antibody; anti-VEGF monoclonal antibody; Avastin; rhuMAb VEGF
Other: laboratory biomarker analysis — Correlative studies
Other: pharmacological study — Correlative studies
  Arms: Phase I Dose Finding; Phase I Dose Finding - Level 1 5mg; Phase I Dose Finding - Level 2 10mg; Phase I Dose Finding - Level 3 20mg

SUMMARY:
This phase I/II trial is studying the side effects and the best dose of RO4929097 to see how well it works when given together with bevacizumab compared to bevacizumab alone in treating patients with progressive or recurrent malignant glioma. RO4929097 may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Monoclonal antibodies, such as bevacizumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Giving RO4929097 together with bevacizumab may kill more tumor cells.

DETAILED DESCRIPTION:
Phase I

Primary Objective:

1. To assess the safety profile of R04929097 in combination with bevacizumab and to determine a recommended Phase II dose of R04929097 in combination with bevacizumab in patients with recurrent malignant glioma

   Secondary Objectives:
2. To describe the toxicity associated with this combination regimen
3. To assess pharmacokinetics of R04929097 in combination with bevacizumab

Phase II I. Assess the safety profile and the recommended phase II dose of gamma-secretase inhibitor RO4929097 (RO4929097) in combination with bevacizumab in patients with recurrent malignant glioma.

II. Assess the progression-free survival at 6 months of patients treated with this regimen.

III. Compare the overall survival of patients with recurrent glioblastoma treated with RO4929097 and bevacizumab versus bevacizumab alone.

SECONDARY OBJECTIVES:

I. Describe the toxicity associated with this regimen in these patients. II. Assess the pharmacokinetics of this regimen in these patients. III. Estimate the proportion of patients alive and progression-free survival at 6 months in patients treated with RO4929097 and bevacizumab versus bevacizumab alone.

IV. Evaluate the safety and tolerability of these regimens in these patients. V. Explore potential prognostic biomarkers from glioma tissue at baseline and potential association with Notch pathway inhibition.

OUTLINE: This is a multicenter, phase I, dose-escalation study of gamma-secretase inhibitor RO4929097 (RO4929097) followed by a randomized phase II study.

PHASE I: Patients receive oral RO4929097 on days 1-3, 8-10, 15-17, and 22-24, and bevacizumab IV over 30-90 minutes on days 1 and 15 (days 2 or 3 and 15 of course 1 only). Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

PHASE II: Patients are randomized* to 1 of 2 treatment arms.

ARM I: Patients receive oral RO4929097 on days 1-3, 8-10, 15-17, and 22-24, and bevacizumab IV over 30-90 minutes on days 1 and 15.

ARM II: Patients receive bevacizumab as in arm I.

In both arms, courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

NOTE: *If phase II single-arm study demonstrates effectiveness, it will proceed to the phase II randomized study.

Some patients undergo blood sample collection for pharmacokinetic studies. Archived tumor tissue samples are analyzed for potential biomarkers and Notch pathway inhibition.

After completion of study therapy, patients are followed up every 2 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed malignant glioma (phase I)

  * Glioblastoma
  * Anaplastic astrocytoma
  * Anaplastic oligodendroglioma
  * Mixed anaplastic oligoastrocytoma
* Histologically confirmed glioblastoma following radiotherapy and temozolomide (phase II)
* Progressive or recurrent disease after conformal external-beam radiation therapy and concurrent temozolomide, followed by ≥ 1 adjuvant course of temozolomide
* Measurable disease by MRI within the past 2 weeks
* Tumor tissue form indicating availability of archived tissue from initial resection at diagnosis of malignant glioma completed and signed by a pathologist
* Karnofsky performance status 60-100%
* ANC ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Hemoglobin ≥ 9 g/dL
* Total bilirubin normal
* AST and ALT ≤ 2.5 times upper limit of normal
* Creatinine normal OR creatinine clearance ≥ 60 mL/min

  * Urine protein: If proteinuria ≥ +2 protein, a protein level should be < 1,000 mg by a 24-hour urine collection
* Electrolytes (calcium, chloride, magnesium, potassium, phosphorus, sodium) within institutional normal limits
* Fertile patients must use 2 forms of effective contraception before, during, and for ≥ 12 months (6 months phase II, bevacizumab arm only) after treatment
* Negative pregnancy test
* Not pregnant or nursing
* At least 5 years since prior malignancy except nonmelanoma skin cancer, or carcinoma in situ of the cervix, breast, or bladder
* Mini Mental State Exam score of ≥ 15
* Must be able to tolerate MRI

Exclusion Criteria:

* No serious concurrent infection or medical illness that would jeopardize the ability of the patient to receive the treatment outline in this protocol with reasonable safety
* No history of allergic reactions attributed to compounds of similar chemical or biological composition to gamma-secretase inhibitor RO4929097 or bevacizumab
* Must be able to swallow capsules
* No malabsorption syndrome or other condition that would interfere with intestinal absorption
* No baseline QTcF > 450 msec (male) or QTcF > 470 msec (female)
* Not history of being serologically positive for hepatitis A, B, or C
* No history of cirrhosis
* No uncontrolled hypocalcemia, hypomagnesemia, hyponatremia, or hypokalemia despite adequate electrolyte supplementation
* No uncontrolled intercurrent illness including, but not limited to, any of the following:

  * Ongoing or active infection
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * A history of torsades de pointes or other significant cardiac arrhythmias other than chronic, stable atrial fibrillation
  * Psychiatric illness and/or social situations that would limit compliance with study requirements
* No serious or non-healing wound, ulcer, or bone fracture
* No history of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within the past 6 months
* No significant vascular disease (e.g., aortic aneurysm requiring surgical repair or recent peripheral arterial thrombosis) within the past 6 months
* No clinically significant cardiovascular disease, including any of the following:

  * Inadequately controlled hypertension (systolic BP > 160 mm Hg and/or diastolic BP > 90 mm Hg) despite antihypertensive medication
  * History of cerebrovascular accident or transient ischemic attack at any time
  * Myocardial infarction or unstable angina within the past 12 months
  * NYHA grade II-IV congestive heart failure
  * Serious and inadequately controlled cardiac arrhythmia
  * Significant vascular disease (e.g., aortic aneurysm or history of aortic dissection)
  * Clinically significant peripheral vascular disease
* No evidence of bleeding diathesis or coagulopathy
* No known hypersensitivity to Chinese hamster ovary cell products or other recombinant human antibodies
* No requirement for antiarrhythmics or other medications known to prolong QTc
* One or 2 prior treatment regimens allowed
* Recovered from severe toxicity of prior therapy
* At least 3 months since prior radiotherapy
* At least 6 weeks since prior nitrosourea
* At least 3 weeks since prior chemotherapy
* At least 4 weeks since prior and no other concurrent investigational agents
* At least 2 weeks since prior non-cytotoxic, FDA-approved agent (e.g., Tarceva [erlotinib hydrochloride], hydroxychloroquine, bevacizumab, etc.)
* At least 28 days since any prior surgery
* No prior γ-secretase inhibitors and/or bevacizumab
* At least 10 days since prior and no concurrent enzyme-inducing anti-epileptic drug
* No concurrent combination antiretroviral therapy for HIV-positive patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2010-12; Primary Completion 2013-01 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edward Pan, MD, Principal Investigator — National Cancer Institute (NCI)
Locations (4):
- United States (4):
  - University of California at Los Angeles (UCLA ), Los Angeles, California
  - University of California San Francisco Medical Center-Parnassus, San Francisco, California
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Memorial Sloan-Kettering Cancer Center, New York, New York

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Phase I trial started 8/2011 and enrollment closed 7/31/12. 13 total patients treated by RO4929097 (5, 10, 20mg/kg) in combo with bevacizumab. 1 treated pt ineligible for study. Analysis data for toxicity included 13 treated pts. Analytical dataset results other than toxicity included 12 eligible pts only. Pts enrolled from outpt medical clinics
Pre-assignment Details: A decision was made from the company, Roche, the owner and developer of RO4929097, that as of 7/31/12 there would be no further supply of RO4929097 and all clinical trials using this drug must stop accruing and treating patients. Hence our ABTC 1002 study was stopped during the phase 1 with 13 pt accrued and the Phase 2 was unable to begin.
Groups:
- Phase I Dose Finding - Level 1 5mg: Patients receive oral gamma-secretase/Notch signalling pathway inhibitor RO49290977 5mg on days 1-3, 8-10, 15-17, and 22-24, and bevacizumab IV over 30-90 minutes on days 1 and 15. Other: blood samples for pharmacological study; archived tumor tissue slides for laboratory biomarker analysis.
  gamma-secretase/Notch signalling pathway inhibitor RO4929097: Given orally
  bevacizumab: Given IV
  laboratory biomarker analysis: Correlative studies
  pharmacological study: Correlative studies
- Phase I Dose Finding Level 2 10mg: Patients receive oral gamma-secretase/Notch signalling pathway inhibitor RO49290977 10mg on days 1-3, 8-10, 15-17, and 22-24, and bevacizumab IV over 30-90 minutes on days 1 and 15. Other: blood samples for pharmacological study; archived tumor tissue slides for laboratory biomarker analysis.
  gamma-secretase/Notch signalling pathway inhibitor RO4929097: Given orally
  bevacizumab: Given IV
  laboratory biomarker analysis: Correlative studies
  pharmacological study: Correlative studies
- Phase I Dose Finding Level 3 20mg: Patients receive oral gamma-secretase/Notch signalling pathway inhibitor RO49290977 20mg on days 1-3, 8-10, 15-17, and 22-24, and bevacizumab IV over 30-90 minutes on days 1 and 15. Other: blood samples for pharmacological study; archived tumor tissue slides for laboratory biomarker analysis.
  gamma-secretase/Notch signalling pathway inhibitor RO4929097: Given orally
  bevacizumab: Given IV
  laboratory biomarker analysis: Correlative studies
  pharmacological study: Correlative studies
Period: Overall Study
Arm/Group | Phase I Dose Finding - Level 1 5mg | Phase I Dose Finding Level 2 10mg | Phase I Dose Finding Level 3 20mg
Started | 4 | 6 | 3
Completed | 4 | 6 | 3
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: 1 pt not eligible for study and hence was not included in the analytical analysis
Groups:
- Phase I Dose Finding: Patients receive oral gamma-secretase/Notch signalling pathway inhibitor RO49290977 on days 1-3, 8-10, 15-17, and 22-24, and bevacizumab IV over 30-90 minutes on days 1 and 15. Other: blood samples for pharmacological study; archived tumor tissue slides for laboratory biomarker analysis.
  gamma-secretase/Notch signalling pathway inhibitor RO4929097: Given orally
  bevacizumab: Given IV
  laboratory biomarker analysis: Correlative studies
  pharmacological study: Correlative studies
Arm/Group | Phase I Dose Finding
Number analyzed (Participants) | 12
Age, Continuous [Median (Full Range); unit: years] | 56 [42 to 62]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 5
Race/Ethnicity, Customized [Number; unit: participants]
  African American | 2
  White | 10
Karnofsky Performance Status [Number; unit: participants] — 100-80: Able to carry on normal activity and to work; No special care needed.
  70-50: Unable to work; able to live at home and care for most personal needs; varying amount of assistance needed.
  40-10: Unable to care for self; Requires equivalent of institutional or hospital care;diseases may be progressing rapidly.
  0: Dead
  participants
    90 | 6
    80 | 5
    70 | 0
    60 | 1
Mini Mental State Examination (MMSE) [Median (Full Range); unit: units on a scale] — Measure of Cognitive impairment
  24-30 No cognitive impairment 18-23 Mild cognitive impairment 0-17 Severe cognitive impairment
  Series of questions with a point value for each question which is summed to give a total final score.
  units on a scale | 29 [21 to 30]
Prior Relapses [Number; unit: participants]
  1 relapse | 8
  2 relapes | 3
  3 relapses | 1
Initial Procedure [Number; unit: participants]
  biopsy | 1
  Resection | 11
Initial Histological Diagnosis [Number; unit: participants]
  Glioblastoma | 10
  Other | 2

OUTCOME MEASURES:

1. Primary Outcome: Maximum-tolerated Dose and the Recommended Phase II Dose of Gamma-secretase Inhibitor RO4929097 in Combination With Bevacizumab Determined by Dose-limiting Toxicity Rate (Phase I)
Description: Pts were treated at escalating dose levels of RO4929097 (Dose levels: 5, 10 or 20 mg) for an observed evaluation at the end of a 4week period. 3 pts treated at each cohort if less than or equal to 33% dose will be escalated. Pts must receive one dose of treatment to be evaluated for toxicity. A standard 3+3 dose escalation method will be used
Time Frame: 28 days
Population: RO4929097 Days 1-3 weekly (doses 5,10, 20 mg) + Bev 10mg/kg IV q2 wks - cycle 28 days. 3+3 dose escalation method will be used. Target DLT is > or equal to 33%
Measure: Number; unit: mg
Arm/Group | Phase I Dose Finding
Number analyzed (Participants) | 13
mg | 10

2. Secondary Outcome: Toxicity Description (Dose Limiting Toxicity-DLT) of Gamma-secretase Inhibitor RO4929097 in Combination With Bevacizumab
Description: Pts were treated at escalating dose levels of RO4929097 (Dose levels: 5, 10 or 20 mg) for an observed evaluation at the end of a 4week period. 3 pts treated at each cohort. Pts must receive one dose of treatment to be evaluated for toxicity. Toxcity description associated with combination of RO4929097 and Bevacizumab
Time Frame: 28 days - 1 cycle
Population: DLT Defintion, must be related to RO and/or Bev: ANC </= 500/μL or second time ANC <1,000/μL; PLTs </= 25,000/μL or second time platelets <50,000/μL; Febrile neutropenia;Thrombocytopenic bleeding (platelets <50,000/μL and with clinically significant bleeding); Delay of treatment > 14 days ;grade 3 or 4 non-hematological toxicity (some exceptions)
Measure: Number; unit: participants
Arm/Group | Phase I Dose Finding - Level 1 5mg | Phase I Dose Finding Level 2 10mg | Phase I Dose Finding Level 3 20mg
Number analyzed (Participants) | 4 | 6 | 3
participants | 0 | 1 | 0

3. Secondary Outcome: Measurement of Cmax to Determine the Effect of Bevacizumab on the Plasma Pharmacokinetics of RO4929097 Day 1
Description: all pts at all dose levels (5,10 and 20mg) will have pks collected. 10 samples will be collected at various time points over a 24 hour time point. Samples will be collected on the first day of treatment during cycle 1.
  For initial cycle (Cycle 1) bevacizumab was not given until 2 or 3 days after all PKs samples of initial dose of RO49290977 was collected
Time Frame: 24 hrs
Population: Day One only
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Groups:
- Phase I Dose Finding - Level 1 5mg: Patients receive oral gamma-secretase/Notch signalling pathway inhibitor RO49290977 5mg on days 1-3, 8-10, 15-17, and 22-24, and bevacizumab IV over 30-90 minutes on days 1 and 15. Other: blood samples for pharmacological study; archived tumor tissue slides for laboratory biomarker analysis.
  For initial cycle (Cycle 1) bevacizumab was not given until 2 or 3 days after all PKs samples of initial dose of RO49290977 was collected
  gamma-secretase/Notch signalling pathway inhibitor RO4929097: Given orally
  bevacizumab: Given IV
  laboratory biomarker analysis: Correlative studies
  pharmacological study: Correlative studies
- Phase I Dose Finding Level 2 10mg: Patients receive oral gamma-secretase/Notch signalling pathway inhibitor RO49290977 10mg on days 1-3, 8-10, 15-17, and 22-24, and bevacizumab IV over 30-90 minutes on days 1 and 15. Other: blood samples for pharmacological study; archived tumor tissue slides for laboratory biomarker analysis.
  For initial cycle (Cycle 1) bevacizumab was not given until 2 or 3 days after all PKs samples of initial dose of RO49290977 was collected
  gamma-secretase/Notch signalling pathway inhibitor RO4929097: Given orally
  bevacizumab: Given IV
  laboratory biomarker analysis: Correlative studies
  pharmacological study: Correlative studies
- Phase I Dose Finding Level 3 20mg: Patients receive oral gamma-secretase/Notch signalling pathway inhibitor RO49290977 20mg on days 1-3, 8-10, 15-17, and 22-24, and bevacizumab IV over 30-90 minutes on days 1 and 15. Other: blood samples for pharmacological study; archived tumor tissue slides for laboratory biomarker analysis.
  For initial cycle (Cycle 1) bevacizumab was not given until 2 or 3 days after all PKs samples of initial dose of RO49290977 was collected
  gamma-secretase/Notch signalling pathway inhibitor RO4929097: Given orally
  bevacizumab: Given IV
  laboratory biomarker analysis: Correlative studies
  pharmacological study: Correlative studies
Arm/Group | Phase I Dose Finding - Level 1 5mg | Phase I Dose Finding Level 2 10mg | Phase I Dose Finding Level 3 20mg
Number analyzed (Participants) | 4 | 6 | 3
ng/mL | 129 (41) | 177 (32) | 241 (172)

4. Secondary Outcome: Measurement of Cmax to Determine the Effect of Bevacizumab on the Plasma Pharmacokinetics of RO4929097 Day 15
Description: all pts at all dose levels (5,10 and 20mg) will have pks collected. 10 samples will be collected at various time points over a 24 hour time point. Samples will be collected on the 15th day of treatment during cycle 1.
Time Frame: 24hr
Population: Day 15 only. Level 2 10mg only had 5pts with evaluable PKs at day 15
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Arm/Group | Phase I Dose Finding - Level 1 5mg | Phase I Dose Finding Level 2 10mg | Phase I Dose Finding Level 3 20mg
Number analyzed (Participants) | 4 | 5 | 3
ng/mL | 117 (37) | 189 (49) | 245 (192)

5. Secondary Outcome: Measurement of AUC24 to Determine the Effect of Bevacizumab on the Plasma Pharmacokinetics of RO4929097 Day 1
Description: all pts at all dose levels (5,10 and 20mg) will have pks collected. 10 samples will be collected at various time points over a 24 hour time point. Samples will be collected on the first day of treatment during cycle 1.
Time Frame: 24hrs
Population: Day 1
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Phase I Dose Finding - Level 1 5mg | Phase I Dose Finding Level 2 10mg | Phase I Dose Finding Level 3 20mg
Number analyzed (Participants) | 4 | 6 | 3
ng*h/mL | 1,215 (361) | 2,385 (606) | 2,232 (781)

6. Secondary Outcome: Measurement of AUC24 to Determine the Effect of Bevacizumab on the Plasma Pharmacokinetics of RO4929097 Day 15
Description: as for outcome 4
Time Frame: 24hr
Population: Day 15. Only 4 pts samples were evaluable for AUC 24 at the10mg dose.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Phase I Dose Finding - Level 1 5mg | Phase I Dose Finding Level 2 10mg | Phase I Dose Finding Level 3 20mg
Number analyzed (Participants) | 4 | 4 | 3
ng*h/mL | 1,212 (355) | 2,351 (1,071) | 2,555 (1,363)

ADVERSE EVENTS:
Time Frame: First dose of drug, than weekly during cycle 1 and then once every 28 days until disease progression, approximately 1 year
Arm/Group | Phase I Dose Finding
Serious Adverse Events (participants affected / at risk) | 1/13
Other Adverse Events (participants affected / at risk) | 13/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I Dose Finding (N=13)
Colonic perforation (Gastrointestinal disorders) | 1 (1)
Sigmoidectomy (Gastrointestinal disorders) | 1 (1)
Platelet count decreased (Investigations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I Dose Finding (N=13)
Alanine aminotransferase increased (Investigations) | 4 (4)
alkaline phosphatase increased (Investigations) | 1 (1)
alopecia (Skin and subcutaneous tissue disorders) | 2 (2)
anemia (Blood and lymphatic system disorders) | 2 (2)
arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
aspartate aminotransferase increase (Investigations) | 3 (3)
blood bilirubin increase (Investigations) | 1 (1)
constipation (Gastrointestinal disorders) | 2 (2)
dyspepsia (Gastrointestinal disorders) | 2 (2)
dyspagia (Gastrointestinal disorders) | 1 (1)
dysphasia (Nervous system disorders) | 1 (1)
cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
edema limbs (General disorders) | 1 (1)
epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
fall (Injury, poisoning and procedural complications) | 2 (2)
fatigue (General disorders) | 7 (7)
headaches (Nervous system disorders) | 3 (3)
hematoma (Vascular disorders) | 1 (1)
hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
hypertension (Vascular disorders) | 5 (5)
hypoalbuminemia (Metabolism and nutrition disorders) | 2 (2)
hypokalemia (Metabolism and nutrition disorders) | 1 (1)
hypomagnesemia (Metabolism and nutrition disorders) | 1 (1)
hypophosphatemia (Metabolism and nutrition disorders) | 2 (2)
irregular menstruation (Reproductive system and breast disorders) | 1 (1)
mucositis oral (Gastrointestinal disorders) | 2 (2)
nausea (Gastrointestinal disorders) | 2 (2)
neutrophil count decrease (Investigations) | 2 (2)
non-cardiac chest pain (General disorders) | 1 (1)
platelet count decrease (Investigations) | 5 (5)
vascular disorder (Cardiac disorders) | 1 (1)
voice alteration (Respiratory, thoracic and mediastinal disorders) | 2 (2)
vomiting (Gastrointestinal disorders) | 1 (1)
white blood cells decrease (Investigations) | 5 (5)

LIMITATIONS AND CAVEATS:
This is Phase 1/Phase 2 Study. It closed prematurely by Roche, study still in Phase 1. Roche halted pt enrollment in ALL clinical trials w/ RO4929097 & cease production of drug & development. Phase 2 of this study was never activated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less